CLINICAL TRIAL: NCT06877780
Title: Patient-reported Outcome Measures of Two Different Treatment Protocols to Manage Growing Patients With Skeletal Class III and Maxillary Constriction: A Randomized Controlled Trial
Brief Title: Evaluation of Pain and Functional Impairments When Treating Class III Malocclusion Using Two Treatment Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-5-2025
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Class III Malocclusion; Maxillary Deficiency
MeSH Terms: conditions — Malocclusion, Angle Class III; Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removable mandibular retractor with slow maxillary expansion (Active Comparator): Patients in this group will undergo treatment using a removable mandibular retractor (RMR) associated with slow maxillary expansion (SME).
  Interventions: Device: RMR with SME
- Bone-anchored intermaxillary traction with rapid maxillary expansion (Experimental): Patients in this group will undergo treatment using bone-anchored intermaxillary traction (BAIMT) associated with rapid maxillary expansion (RME).
  Interventions: Device: BAIMT with RME

INTERVENTIONS:
Device: RMR with SME — The RMR will be used in conjunction with slow maxillary expansion
  Arms: Removable mandibular retractor with slow maxillary expansion
Device: BAIMT with RME — The bone-anchored intermaxillary traction will be used with rapid maxillary expansion
  Arms: Bone-anchored intermaxillary traction with rapid maxillary expansion

SUMMARY:
A clinical examination of each recalled candidate patient will be carried out at Adib Al Lahham Centre at the Ministry of Health Damascus to ensure that he/she meets the inclusion criteria. Following obtaining the full records, including a lateral cephalometric radiograph, additional checking will be made to classify the skeletal relationship (class III relationship) of each possible candidate for this work.

This trial compares two groups of patients who suffered from Class III malocclusion associated with maxillary constriction.

Experimental Group: Patients in this group will undergo treatment using bone-anchored intermaxillary traction (BAIMT) associated with rapid maxillary expansion (RME).

Control Group: Patients in this group will undergo treatment using a removable mandibular retractor (RMR) associated with slow maxillary expansion (SME).

DETAILED DESCRIPTION:
Treating skeletal Class III malocclusion presents challenges. However, various methods have been implemented for treating Class III cases through growth modification during the primary and mixed dentition stages, such as the removable mandibular retractor (RMR) and recently bone-anchored intermaxillary traction (BAIMT) system. In orthodontics, there has been increasing interest in assessing patient-reported outcome measures (PROMs) for two reasons: First, the patient's psychosocial well-being enhances collaboration during treatment. Second, the results of orthodontic treatment may advance if the patient is informed and self-assured regarding their treatment.

Participants will be chosen from patients attending the Adib Al Lahham Centre at the Ministry of Health Damascus. Eligible patients with Class III malocclusion associated with maxillary constriction who meet the inclusion criteria will be asked to participate in this study following a screening conducted by the researcher. Informed consent will be acquired from all patients who consent to participate in the survey after receiving an information sheet.

For BAIMT with the RME group, a modified Hyrax palatal expander with posterior bite planes will be bonded. The expander will also have hooks welded distal to the first molars to attach elastic bands. Two self-drilling mini screws will be inserted buccally between the roots of the mandibular canine and the first premolar. Then, intermaxillary elastics will be placed between the hooks and the mandibular.

FOR RMR with SME group, patients in this group will be provided with an RMR appliance containing a midline split that included an expansion screw, and an anterior sagittal expansion screw which will be utilized when necessary to rectify the upper incisors axes.

A change in the relationship of the incisor from a negative overjet to a positive one (i.e., + 1.5 mm or greater) will be deemed a sign of successful treatment in the sagittal plane. If the defect in the transverse plane is addressed first, the expansion will be halted, and the patient will be asked to keep wearing the appliance until the deficiency in the sagittal plane is corrected. On the other hand, if the defect in the sagittal plane is corrected initially, the process will be reversed.

The levels of pain, functional impairment, and confidence will be self-reported using a questionnaire with a 4-point Likert scale administered at five evaluation times during the ﬁrst 6 months of treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Growing patients between the ages of 12-15 of either gender.
* Angle's class III malocclusion.
* Skeletal class III (-4 < ANB < + 1).
* Anterior crossbite involving two or more teeth or edge-to-edge incisor relationship with or without a forward shift of the mandible during closure.
* The incisor mandibular plane's (IMPA) angle should be between 85° and 100°.
* Maxillary constriction necessitates expansion.

Exclusion Criteria:

* Skeletal class III malocclusion is mainly caused by maxillary retrognathism.
* Severe skeletal class III, mainly resulting from mandibular prognathism.
* Contraindications for the application of the mini-screws.
* The presence of supernumerary teeth or missing ones except for the third molars.
* The presence of cleft lip or craniofacial syndromes and/or palate abnormalities.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in the feeling of pressure at the soft tissues | The questionnaire will be distributed to the patients at five assessment times: (T1) one day after the active treatment initiation, (T2) after one week (T3) after a month, (T4) after 3 months, and (T5) after 6 months of treatment initiation.
  Patients will be asked to identify their pressure at the soft tissues by asking, " Do you suffer from pressure at the soft tissues while wearing the device/applying the elastics?" They will choose their possible answer from one of the following options according to the four-point scale: (1) None (2) mild (3) moderate (4) severe, which corresponds to the following numbers (0-1-2-3).
Change in the perception of pain | The questionnaire will be distributed to the patients at five assessment times: (T1) one day after the active treatment initiation, (T2) after one week (T3) after a month, (T4) after 3 months, and (T5) after 6 months of treatment initiation.
  Patients will be asked to identify their pain perception by answering, " Do you suffer from pain while wearing the device/applying the elastics?" They will choose their possible answer from one of the following options according to the four-point scale: (1) None (2) mild (3) moderate (4) severe, which corresponds to the following numbers (0-1-2-3).

SECONDARY OUTCOMES:
Change in speech difficulties | The questionnaire will be distributed to the patients at five assessment times: (T1) one day after the active treatment initiation, (T2) after one week (T3) after a month, (T4) after 3 months, and (T5) after 6 months of treatment initiation.
  Patients will be asked to identify their perception of speech difficulties by answering, " Do you suffer from speech difficulties while wearing the device/applying the elastics?" They will choose their possible answer from one of the following options according to the four-point scale: (1) None (2) mild (3) moderate (4) severe, which corresponds to the following numbers (0-1-2-3).
Change in the swallowing difficulties | The questionnaire will be distributed to the patients at five assessment times: (T1) one day after the active treatment initiation, (T2) after one week (T3) after a month, (T4) after 3 months, and (T5) after 6 months of treatment initiation.
  Patients will be asked to identify their perception of swallowing disability by answering, " Do you suffer from a swallowing disability while wearing the device/applying the elastics?" They will choose their possible answer from one of the following options according to the four-point scale: (1) None (2) mild (3) moderate (4) severe, which corresponds to the following numbers (0-1-2-3).
Change in the limitation in the movement of the mandible. | The questionnaire will be distributed to the patients at five assessment times: (T1) one day after the active treatment initiation, (T2) after one week (T3) after a month, (T4) after 3 months, and (T5) after 6 months of treatment initiation.
  Patients will be asked to identify their perception of limitation in the movement of the mandible by answering, "Do you suffer from a limitation in the movement of the mandible while wearing the device/applying the elastics?" They will choose their possible answer from one of the following options according to the four-point scale: (1) None (2) mild (3) moderate (4) severe, which corresponds to the following numbers (0-1-2-3)
Change in the feeling of embarrassment | The questionnaire will be distributed to the patients at five assessment times: (T1) one day after the active treatment initiation, (T2) after one week (T3) after a month, (T4) after 3 months, and (T5) after 6 months of treatment initiation.
  Patients will be asked to identify their shame by asking, " Do you feel ashamed while wearing the device/applying the elastics?" They will choose their possible answer from one of the following options according to the four-point scale: (1) None (2) mild (3) moderate (4) severe, which corresponds to the following numbers (0-1-2-3).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S. Zakaria, DDS MSc, Principal Investigator — Department of Orthodontics, School of Dental Sciences, USM Health Campus, Kelantan, Malaysia; Rozita Hassan, DDS MSc PhD, Study Chair — Department of Orthodontics, School of Dental Sciences, USM Health Campus, Kelantan, Malaysia
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abed Al Jawad FH, Alhashimi NA. Evaluation of self-perceived pain and jaw function impairment in children undergoing slow and rapid maxillary expansion. Angle Orthod. 2021 Nov 1;91(6):725-732. doi: 10.2319/020221-100.1. PMID 34033675
- [Background] Rabah N, Al-Ibrahim HM, Hajeer MY, Ajaj MA, Mahmoud G. Assessment of Patient-Centered Outcomes When Treating Maxillary Constriction Using a Slow Removable Versus a Rapid Fixed Expansion Appliance in the Adolescence Period: A Randomized Controlled Trial. Cureus. 2022 Mar 3;14(3):e22793. doi: 10.7759/cureus.22793. eCollection 2022 Mar. PMID 35261839
- [Background] Saleh M, Hajeer MY, Al-Jundi A. Assessment of pain and discomfort during early orthodontic treatment of skeletal Class III malocclusion using the Removable Mandibular Retractor Appliance. Eur J Paediatr Dent. 2013 Jun;14(2):119-24. PMID 23758461
- [Background] Ryan FS, Cunningham SJ. Patient-reported outcome measures and orthodontics. J Orthod. 2018 Jun;45(2):63-64. doi: 10.1080/14653125.2018.1472729. No abstract available. PMID 29857794
- [Background] Sergl HG, Zentner A. A comparative assessment of acceptance of different types of functional appliances. Eur J Orthod. 1998 Oct;20(5):517-24. doi: 10.1093/ejo/20.5.517. PMID 9825554
- [Derived] Zakaria AS, Hassan R, Baharin F, Alfailany DT, Hajeer MY, Al-Hamod IA, Al-Sabbagh R. Evaluation of Patient-reported Outcome Measures during the Correction of Skeletal Class III Malocclusion with Maxillary Constriction in Early Adolescence. J Contemp Dent Pract. 2025 Jun 1;26(6):598-607. doi: 10.5005/jp-journals-10024-3901. PMID 41040030